CLINICAL TRIAL: NCT07139795
Title: The Mind-Body Project
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northeastern University (Other)
Responsible Party: Principal Investigator, Neha Gothe, Associate Professor, Northeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB:25-06-24
Record Dates: First submitted 2025-08-15; First posted 2025-08-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will engage in group mindful eating sessions 1x/week for 75 minutes. Participants will be encouraged to attend at least 2x/week, 45-minute yoga sessions.
  Interventions: Behavioral: Mindful eating and movement
- Waitlist Control (No Intervention): Participants assigned to the waitlist control group will complete all baseline and follow-up assessments at the same time as the intervention group. They will receive the same 8-week program after the completion of all assessments by all participants.

INTERVENTIONS:
Behavioral: Mindful eating and movement — Group mindful eating sessions will be conducted once per week, one hour per session, for eight weeks. Participants will be encouraged to attend at least two, 45-minute yoga sessions per week.
  Arms: Intervention Group

SUMMARY:
The goal of this pilot clinical trial is to learn if a combined mindful eating and mindful movement (yoga) program is feasible and acceptable for people with overweight/obesity. The main questions it aims to answer are:

1. What is the feasibility and acceptability of an 8-week mindful eating and yoga intervention for adults with overweight/obesity?
2. Does the program bring about changes in mindfulness, dietary behaviors, and physical activity?
3. Does the program lead to positive changes in body composition, and key biomarkers of blood sugar and lipids assessed via a blood panel using a finger stick procedure (no venous blood draw).

Researchers will compare the 8-week mindful eating and movement intervention to a waitlist control group.

Participants will:

Be assigned to the 8-week intervention or waitlist group. Participate 2x/week in the mindful eating and movement sessions. Complete assessments of feasibility and acceptability as well as self-report and objective assessments describe above.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Body Mass Index (BMI) > 27 kg/m2
* Ambulatory
* Ability to read, write, and understand English
* Intention to remain in the Boston area for the duration of the study
* Good or corrected vision and hearing
* Not currently enrolled in a physical activity or nutrition study
* Affiliated with Northeastern as a student, faculty, staff, or alumni
* No participation in a weight loss study in the past 12 months
* Willingness to participate in all study measurements and activities of their assigned group
* Ability to provide informed consent
* No bariatric surgery in the past five years or plans for bariatric surgery within the study period

Exclusion Criteria:

* < 18 years of age
* BMI < 27 kg/m2
* Non-ambulatory (i.e., use of walkers, wheelchairs)
* Participation in a weight loss study in the past 12 months
* Currently enrolled in a different physical activity or nutrition study
* Significant problems with vision or hearing
* Unwilling to participate in all study measurements and/or activities of their assigned group
* Participation in guided yoga sessions in the past three months
* Adults not affiliated with Northeastern as a student, faculty, staff, or alumni
* Current cancer diagnosis and going through active treatment (chemotherapy, radiation)
* Pregnant, breastfeeding, or plans to become pregnant during the three-month intervention
* Inability to provide informed consent
* Bariatric surgery within the past five years or plans for bariatric surgery within the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Primary endpoint: 8-weeks
  Defined as achieving the target recruitment sample in a 12-month period, 80% retention, 70% attendance rate, and no serious adverse events.
Acceptability | Primary endpoint: 8-weeks
  Defined as >5/7 on acceptability questionnaire (1 = unacceptable, 7 = very acceptable)

CONTACTS AND LOCATIONS:
Overall Officials: Neha P Gothe, PhD, MA, MS, Principal Investigator — Northeastern University
Locations (1):
- Northeastern University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No